CLINICAL TRIAL: NCT03258203
Title: Obesity Genes, Energy Regulation in Response to Weight-Loss
Brief Title: Gene-Environment Interaction and Precision Nutrition on Adiposity, Glycemic, Lipids Changes, and Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lu Qi, Director of Tulane University Obesity Research Center, Tulane University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01DK091718 (NIH)
Record Dates: First submitted 2017-08-11; First posted 2017-08-23 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- diet 1 (Experimental): diet with moderate in fat (40% energy) and protein(15%)
  Interventions: Other: Preventing Overweight Using Novel Dietary Strategies
- diet 2 (Experimental): diet with moderate in fat (40% energy) and protein(25%)
  Interventions: Other: Preventing Overweight Using Novel Dietary Strategies
- diet 3 (Experimental): diet with low in fat (20% energy) and protein(15%)
  Interventions: Other: Preventing Overweight Using Novel Dietary Strategies
- diet 4 (Experimental): diet with low in fat (20% energy) and protein(25%)
  Interventions: Other: Preventing Overweight Using Novel Dietary Strategies

INTERVENTIONS:
Other: Preventing Overweight Using Novel Dietary Strategies — The study tests the effectiveness for weight loss and weight maintenance of four diets differing in macronutrient composition: moderate in fat (40% energy) with two different protein levels (15% and 25%), and low in fat (20% energy), also with 15% and 25% protein levels.

SUMMARY:
The purpose of this study is to test the interactions between the genes and diet interventions varying in macronutrient intake on glycemic, waist circumference, body weight, visceral fat and lipids changes. In the POUNDS LOST, all of the 811 participants DNA was extracted from the buffy coat fraction of centrifuged blood using the QIAmp blood kit (Qiagen, Chatsworth, CA). Single nucleotide polymorphisms were genotyped using the OpenArray™ SNP genotyping system (BioTrove, Woburn, MA). The study is only accepting participants in the Boston, Massachusetts or Baton Rouge, Louisiana area. For further enrollment information in Boston or Baton Rouge, see Eligibility Criteria or Design Narrative.

Besides, the investigators integrated novel pathway analyses in large cohorts and comprehensive genetic analyses on long-term weight loss and mechanisms in randomized diet intervention trials would provide very important evidence to unravel the etiology of obesity, and have significant public health and clinical implications. Establishing relationship between genetic variants and diets in determining weight change will help identify individuals at high risk for obesity especially when adherent to specific diet.

DETAILED DESCRIPTION:
The epidemic of obesity has become a major public health problem. Obesity is a multifactorial abnormality that has a genetic basis but requires environmental influences to manifest. Common-form obesity is underpinned by both environmental and genetic factors. Recent genome-wide association studies have identified several genes convincingly related to obesity risk. Testing gene-environment interaction is a relatively new field. Evidence from association studies and intervention trials continues to mount, indicating that genetic components may modify lifestyle effects on the development of obesity. However, these findings are at most preliminary. The interplay between genetic and environmental components may facilitate the choice of more effective and specific measures for obesity prevention based on personalized genetic make-up.

The investigators aimed to examine whether the genetic variation affected glycemic, waist circumference, body weight, visceral fat and lipids changes in response to weight-loss dietary intervention varying in macronutrient intake (target percentages of energy derived from fat, protein, and carbohydrate in the 4 diets were as follows 20%, 15% and 65%; 20%, 25%, and 55%; 40%, 15%, and 45%; and 40%, 25%, and 35%).

The primary outcome is to test the interactions between the genes and diet interventions varying in macronutrient intake on body weight changes. The secondary outcome is to test the interactions between the genes and diet interventions varying in macronutrient intake on glycemic, waist circumference, visceral fat, and lipids changes. Understanding gene-diet interactions in relation to weight loss hold great promise for delivering more efficient prevention and treatment on obesity and related metabolic disorders.

In addition, besides gene-diet interactions, the investigators will also conduct other precision nutrition analysis. These analyses include interactions between pretreatment factors with diet intervention adiposity traits, initial changes induced by diet intervention with various outcomes measured in POUNDS Lost, including body weight, waist circumference, body composition, ectopic fat, and bone health.

ELIGIBILITY:
Inclusion Criteria:

* Only accepting participants in the Boston, Massachusetts or Baton Rouge, Louisiana area
* Between the ages of 30 - 70
* Willing to modify eating pattern according to instructions
* Overweight or obese and in good health with a BMI of 25-40
* Committed to a long-term weight loss and maintenance program
* Willing to attend multiple weight loss group sessions
* Willing to increase activity level

Exclusion Criteria:

* Pregnant, planning to become pregnant, or are breastfeeding
* Unwilling to participate in the schedule of group sessions and individual visits
* Unstable or recent onset of heart disease or any other serious illness
* Cannot change diet due to medical or other reasons
* Planning to leave the area prior to the anticipated end of participation
* Current participation in another clinical trial with an intervention that affects weight change
* Have diabetes that is treated with insulin or hypoglycemic oral medicines
* Diagnosis of psychiatric or emotional problems within 6 months of study
* Currently have an eating disorder
* Have hypothyroidism
* Have an unstable weight

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Test the interactions between the genes and diet interventions varying in macronutrient intake on body weight changes(weight in kilograms) . | measured at Year 2

SECONDARY OUTCOMES:
Test the interactions between the genes and diet interventions varying in macronutrient intake on glycemic changes (mg/dL for fasting glucose,uU/mL for fasting insulin). | measured at Year 2
Test the interactions between the genes and diet interventions varying in macronutrient intake on waist circumference changes (cm). | measured at Year 2
Test the interactions between the genes and diet interventions varying in macronutrient intake on visceral fat changes (%). | measured at Year 2
Test the interactions between the genes and diet interventions varying in macronutrient intake on lipids changes (mg/dL for Total cholesterol, HDL cholesterol, LDL cholesterol and Triglycerides). | measured at Year 2
Test the interactions between the genes and diet interventions varying in macronutrient intake on bone health (Bone mineral density at different skeletal sites). | measured at Year 2
  Bone mineral density was measured by dual-energy X-ray (DEXA)

OTHER OUTCOMES:
Ectopic fat | 2 year (measured at baseline, 6 months, and 2 years)
  Computed tomography (CT) measured hepatic fat, abdominal fat distribution (includes visercal adipose tissue, subcutaneous adipose tissue, and total adipose tissue)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou T, Sun D, Heianza Y, Li X, Champagne CM, LeBoff MS, Shang X, Pei X, Bray GA, Sacks FM, Qi L. Genetically determined vitamin D levels and change in bone density during a weight-loss diet intervention: the Preventing Overweight Using Novel Dietary Strategies (POUNDS Lost) Trial. Am J Clin Nutr. 2018 Nov 1;108(5):1129-1134. doi: 10.1093/ajcn/nqy197. PMID 30475961
- [Derived] Han L, Ma W, Sun D, Heianza Y, Wang T, Zheng Y, Huang T, Duan D, Bray JGA, Champagne CM, Sacks FM, Qi L. Genetic variation of habitual coffee consumption and glycemic changes in response to weight-loss diet intervention: the Preventing Overweight Using Novel Dietary Strategies (POUNDS LOST) trial. Am J Clin Nutr. 2017 Nov;106(5):1321-1326. doi: 10.3945/ajcn.117.156232. Epub 2017 Sep 20. PMID 28931532

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03258203/Prot_SAP_001.pdf